CLINICAL TRIAL: NCT02389712
Title: 16-week Open Randomized Comparative Effectiveness Trial of Lamotrigine vs. Fluoxetine for Bipolar Depression: Pharmacogenomic and Biomarker Predictors of Response
Brief Title: 16-week Comparative Effectiveness Trial of Lamotrigine vs. Fluoxetine for Bipolar Depression
Acronym: FLAME
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulties with recruitment
Sponsor: Mayo Clinic (Other)
Collaborators: J Willard and Alice S. Marriott Foundation (Unknown)
Responsible Party: Principal Investigator, Mark Frye, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-003545-1; UL1TR000135 (NIH)
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Results first posted 2019-06-11 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Mayo Clinic
MeSH Terms: conditions — Bipolar Disorder | interventions — Lamotrigine; Fluoxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lamotrigine (Active Comparator): Subjects on this arm will be randomized to Lamotrigine.
  Interventions: Drug: Lamotrigine
- Fluoxetine (Active Comparator): Subjects on this arm will be randomized to Fluoxetine.
  Interventions: Drug: Fluoxetine

INTERVENTIONS:
Drug: Lamotrigine — Lamotrigine dosing: 25 mg daily x 2 weeks, 50 mg daily x 2 weeks, 100 mg daily x 2 weeks, 200 mg (100 mg bid)) x 4 weeks. If patient still has at least mild depressive symptoms, the dose can be increased to 300 mg daily for 2 weeks and 400 mg for 4 weeks. Dose will be held for treatment response and can be reduced for side effects.
  Other Names: Lamictal
  Arms: Lamotrigine
Drug: Fluoxetine — Fluoxetine dosing: 20mg for month 1, 40mg for month 2, and if still depressed (CGI ≥ 3) 60mg for month 3 and 4. Lower doses of fluoxetine will be prescribed for those with side effects. For known Cytochrome P450 2D6 poor metabolizers, fluoxetine will not be dosed > 40mg.
  Other Names: Prozac
  Arms: Fluoxetine

SUMMARY:
The FLAME Study is a 16-week clinical trial to study treatment with lamotrigine or fluoxetine in bipolar I, II and bipolar schizoaffective depressed adults. The purpose of the trial is to have a better understanding of whether individuals with a particular gene type and other inherited biological markers will have a good response to fluoxetine or lamotrigine, or alternatively, would be more likely to have side effects to this medication.

DETAILED DESCRIPTION:
Depression is the predominant prevailing mood state of bipolar disorder and it is associated with substantial morbidity and mortality. However, in comparison to acute mania, bipolar depression is understudied both from the standpoint of its pathophysiology as well as clinical trials and treatment development. Given the lack of evidence-based guidelines, clinicians and participants enter a treatment phase with little guidance.

The FLAME Study is a 16-week, open randomized comparative effectiveness trial evaluating genomic predictors and biomarkers of response and adverse events to treatment with lamotrigine (n=200) and fluoxetine (n=200) for bipolar I, II and bipolar schizoaffective depressed adults (18-65). Participants will be recruited over a 5-year period.

It is known that functionally significant genetic polymorphisms of pharmacokinetics and pharmacodynamic pathways can influence individual differences in repose to specific medications. We propose to evaluate the contribution of these pharmacogenomic variations to lamotrigine and fluoxetine treatment response and adverse events. We will correlate clinical phenotypes of response and adverse events to treatment with genotype and haplotype variations of drug metabolism, neurotransmitter biosynthesis, (metabolism, storage, release, reuptake), receptor and intracellular signaling-that have been previously implicated to either lamotrigine or fluoxetine. These initial steps will be complemented with genome-wide analysis (GWA), pathway analysis and other candidate gene studies.

Based on our results we aim to develop a translational treatment algorithm of bipolar depression that may help individualized treatment for bipolar depression. This algorithm for participants could potentially increase the likelihood of successful treatment interventions, deliver the "right treatment, for the right participant at the right time", and decrease the number of ineffective treatments and/or risk for serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, age 18-65.
* Outpatients or inpatients with a diagnosis of bipolar I, II or schizoaffective bipolar disorder, depressed phase, non-psychotic, (DSM-5 criteria, Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders Module D confirmed)
* At least mild symptom severity of depression as defined by the Clinical Global Impression for Bipolar Disorder (CGI-BP, Spearing et al. 1997) >2.
* Bipolar I participants must be on conventional mood stabilizing treatment [lithium, divalproex or valproate, or an atypical antipsychotic]. Participants with a bipolar II disorder may pursue the FLAME Study as monotherapy.
* Negative urine pregnancy test.
* Participants not planning pregnancy in the near future (6 months).
* Negative urine toxicology screen (except cannabis).
* No evidence of clinically significant laboratory screening tests (complete blood count (CBC); electrolytes; thyroid stimulating hormone (TSH); creatinine/blood urea nitrogen, Aspartate Aminotransferase (AST)/ALT). Clinical laboratory evaluation within the last three months is acceptable.

Exclusion Criteria:

* Inability or unwilling to provide informed consent.
* Inability to understand English.
* Actively suicidal participants at screening or enrollment visit as defined by a response of 3 or 4 on question 4 of the Bipolar Inventory of Symptoms Scale (BISS).
* Active delusions or hallucinations defined as a score of 3 or 4 on the BISS question 40 (persecutory ideas) or 41 (delusions or hallucinations).
* Impaired insight as defined as a score of 3 or 4 on BISS question 42 (insight).
* Hypomania defined by a BISS manic subscore of ≥15.
* Axis I or II comorbidity that by referring mental health professional and/or study psychiatrist is primary need of treatment. (This will be assessed by the site principal investigator, who has >10 years clinical experience with this population. Hospital discharge summaries and outpatient medical records may be reviewed (i.e., adequate trials of mood stabilizing treatments with minimal to no response, prominent self-injurious behavior in the absence of significant mood symptomatology, or atypical cycle patterns) to make this decision.
* Pregnant participants
* Unwilling or unable to taper any current antidepressant therapy
* Participants currently breastfeeding
* Female not practicing a reliable form of birth control (condom, intrauterine device (IUD), Depo-Provera injection)
* Due to lamotrigine pharmacokinetics, female subjects wishing to commence oral contraceptive therapy (OCT) within 3 months of enrollment date or anticipate discontinuing OCT during study (stable oral contraceptive therapy exception).
* History of active substance abuse disorder within the last 3 months (other than caffeine or cannabis)
* Participants with medical contraindications that preclude lamotrigine or fluoxetine treatment
* History of severe adverse reaction to lamotrigine and/or fluoxetine
* Current carbamazepine or oxcarbazepine treatment
* Unstable active medical illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-03; Primary Completion 2018-05-23 (Actual); Study Completion 2018-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Frye, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lamotrigine | Fluoxetine
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lamotrigine | Fluoxetine | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 27 [27 to 27] | 27 [27 to 27] | 27 [27 to 27]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Inventory for Depressive Symptoms
Time Frame: 12 weeks
Population: Study was terminated due to difficulties with recruitment
Arm/Group | Lamotrigine | Fluoxetine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to week 16 week for both subjects.
Arm/Group | Lamotrigine | Fluoxetine
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT02389712/Prot_SAP_000.pdf